CLINICAL TRIAL: NCT02138630
Title: The Physiological Effects of Capsaicinoid Ingestion on Human Metabolism and Exercise Performance
Brief Title: Capsaicinoid Ingestion, Human Metabolism and Exercise (Phase 2)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Project abandoned
Sponsor: University of Prince Edward Island (Other)
Collaborators: OmniActive Health Technologies (Industry)
Responsible Party: Principal Investigator, Dr. Jamie Burr, Assistant Professor, University of Prince Edward Island
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: OAHTCAPX-003-2014-2
Record Dates: First submitted 2014-05-08; First posted 2014-05-14 (Estimated); Last update posted 2022-06-22 (Actual); Status verified 2015-09

CONDITIONS: Metabolism; Exercise
Keywords: Exercise
MeSH Terms: conditions — Motor Activity | interventions — Capsaicin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Capsaicin (Experimental): Single Capsule, "Capsimax" 100 mg, ingested 60 min prior to exercise
  Interventions: Dietary Supplement: Capsaicin

INTERVENTIONS:
Dietary Supplement: Capsaicin
  Other Names: Capsimax
  Arms: Capsaicin
Dietary Supplement: Placebo — Sugar capsule
  Arms: Placebo

SUMMARY:
Capsaicinoids (the active ingredient in hot peppers) have been shown to cause a moderate increase in energy expenditure (50 kcal/day) as well as reductions in appetite, energy intake, and (visceral) adiposity. As such, there is considerable interest in capsaicinoid for weight loss supplements. Owing to the fact that these changes are believed to be driven by catecholamine release and alterations in fat oxidation, there is growing belief that capsaicin may also offer potential ergogenic benefits (performance enhancement) during exercise, similar to the affect of caffeine, which works through similar pathways. Of particular interest are the recent findings that free-fatty acids in the blood are elevated 2-2.5hrs post ingestion, yet changes in typical cardiovascular or sympathetic nervous tone indicators (heart rate, blood pressure) were unaffected, suggesting some of the negative consequences of other stimulants may be avoided. At present, however, more in depth investigations of the effects on endothelial function, vascular autonomic tone and inflammation are lacking.

Although there are some indications that capsaicinoid ingestion may alter factors associated exercise performance (such as increased fat oxidation for glucose sparing), to date these studies have primarily used very low exercise intensities wherein these effects are typically unnecessary, and results are not generalizable to the typical race intensities of endurance sport competition. Performance measures have also been a noticeably absent outcome from research to date.

Hypotheses: 1), Exercise performance will improve, at a level similar to those demonstrated for caffeine ingestion 2) ratings of perceived exertion will go down with the effect of causing intensity to go up 3) During sustained aerobic activity approaching the aerobic threshold alterations in substrate use will be minimal (but possibly meaningful in regard to performance); alterations at rest will be more pronounced. 4) acute alterations (6o min post single dose) in blood pressure, HRV, arterial stiffness and RMR will mirror the effects observed for more prolonged exposure in phase 1.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be male or female, 18 yr -45yr and free from any known or suspected chronic conditions. General health and suitability to participate in an exercise/health research study will be confirmed through use of the PAR-Q+ screening questionnaire

Exclusion Criteria:

Any participant who has a positive answer to a screening question will be required to seek physician approval prior to any physical exercise. Baseline arrhythmia (tachycardia (>100pbm) and systolic or diastolic hypertension (>140/90 mmHg) will also be reason for exclusion. During baseline anthropometric assessment we will confirm that participants all fall within a typical BMI range (20-30 kg/m2) of either "normal" weight or "overweight", but not "underweight" or "obese". Persons who take cardiovascular medications, metabolic medications, smoke cigarettes, excessively consume alcohol, are prone to heartburn, or have a previous diagnosis of hyperlipidemia or hyperinsulemia will also be excluded

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-06; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Performance | 2 to 4 hours
  Exercise: Time to exhaustion on a cycle ergometer at controlled relative intensity

SECONDARY OUTCOMES:
Substrate Use | 2 to 4 hours
  Measurement of expired gases

CONTACTS AND LOCATIONS:
Locations (1):
- UPEI, Charlottetown, Prince Edward Island, Canada